CLINICAL TRIAL: NCT03207776
Title: A Cluster Randomized, Stepped-Wedge Evaluation of Post Discharge Utilization Among Patients With an Acute Exacerbation of Chronic Obstructive Pulmonary Disorder (COPD)
Brief Title: An Evaluation of Post Discharge Utilization Among Patients With an Acute Exacerbation of COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 00021790
Record Dates: First submitted 2017-06-28; First posted 2017-07-05 (Actual); Results first posted 2019-10-14 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2020-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Treatment of patients in the usual manner based on their diagnosis and resources available at that site (Usual Care).
  Interventions: Other: Usual Care
- Intervention (Other): A group of 4 Usual Care components that are applied consistently and completely amongst all patients who present with COPD acute exacerbation symptoms, plus access to navigator services (COPD Clinical Pathway).
  Interventions: Other: COPD Clinical Pathway

INTERVENTIONS:
Other: Usual Care — Treatment of patients in the usual manner based on their diagnosis and resources available at that site.
  Arms: Control
Other: COPD Clinical Pathway — A group of 4 Usual Care components that are applied consistently and completely amongst all patients who present with COPD acute exacerbation symptoms, plus access to navigator services.
  Arms: Intervention

SUMMARY:
Patients who are hospitalized at select Carolinas Healthcare System (CHS) sites with Chronic Obstructive Pulmonary Disorder (COPD) acute exacerbation symptoms will be treated per the CHS COPD Clinical Pathway. Patient outcomes will be followed, including but not limited to readmission. Patients on the pathway will also have access to navigator services.

DETAILED DESCRIPTION:
Patients hospitalized at participating CHS sites with COPD acute exacerbation symptoms, will be treated per the CHS COPD clinical pathway. The COPD clinical pathway will include four components: (i) discrete, evidence-based care steps (ii) patient navigation, (iii) daily data driven care gap identification, (iv) monthly leadership huddles. These components are all part of usual care for patients in this population, but each component is not applied to patients consistently across the System. For this reason, the pathway will be applied consistently and completely in patients meeting COPD acute exacerbation criteria at participating sites. Patients will be followed for 60 days in total after discharge from their COPD acute exacerbation symptoms to determine the potential effectiveness of complete implementation of all 4 components in the care of COPD patients. Patients on the pathway will also have access to navigator services.

ELIGIBILITY:
Inclusion Criteria:

* Identified as having an acute exacerbation of COPD within 24 hours of admission

Exclusion Criteria:

* Death during the index encounter
* No initial discharge as of the end of the study period

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4832 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2018-02-12 (Actual); Study Completion 2018-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Howard, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (8):
- United States (8):
  - Carolinas Medical Center, Charlotte, North Carolina
  - Carolinas Healthcare System - Pineville, Charlotte, North Carolina
  - Carolinas Healthcare System - University, Charlotte, North Carolina
  - Carolinas Healthcare System - NorthEast, Concord, North Carolina
  - Carolinas Healthcare System - Kings Mountain, Kings Mountain, North Carolina
  - Carolinas Healthcare System Lincoln, Lincolnton, North Carolina
  - Carolinas Healthcare System - Union, Monroe, North Carolina
  - Carolinas Healthcare System - Cleveland, Shelby, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Intervention
Started (All patients with the diagnosis were to receive the intervention) | 2479 | 2353
Completed | 2479 | 2353
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 2479 | 2353 | 4832
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (11.5) | 66.8 (11.0) | 67.3 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1360 | 1366 | 2726
  Male | 1119 | 987 | 2106
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 3 | 8
  Asian | 9 | 3 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 535 | 375 | 910
  White | 1885 | 1928 | 3813
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 45 | 43 | 88
Region of Enrollment [Number; unit: participants]
  United States | 2479 | 2353 | 4832

OUTCOME MEASURES:

1. Primary Outcome: Healthcare Utilization
Description: Occurrence of Emergency Department, inpatient, or observation encounters after the initial encounter at accrual
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 2479 | 2353
Participants | 1080 | 920
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority; p = 0.041, Mixed Models Analysis; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.64 to 0.99]

2. Secondary Outcome: Quality, Comfort, and Care (QCC) Defined Readmission Rate
Description: Readmission to the same facility
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 2479 | 2353
Participants | 321 | 286
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority; p = 0.952, Mixed Models Analysis; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.69 to 1.42]

3. Secondary Outcome: Patient-centric (Protocol Defined) Readmission Rate
Description: Readmission to any facility within Carolinas HealthCare System
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 2479 | 2353
Participants | 753 | 659
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority; p = 0.472, Mixed Models Analysis; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.71 to 1.17]

4. Secondary Outcome: 30-day COPD Specific, Acute Care Utilization to Any Hospital Within the System
Time Frame: 30 day
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 2479 | 2353
Participants | 240 | 179
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority; p = 0.544, Mixed Models Analysis; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.74 to 1.77]

ADVERSE EVENTS:
Time Frame: We followed each patient for 90 days after the hospital discharge
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/2479 | 0/2353
Serious Adverse Events (participants affected / at risk) | 0/2479 | 0/2353
Other Adverse Events (participants affected / at risk) | 0/2479 | 0/2353

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-15): https://cdn.clinicaltrials.gov/large-docs/76/NCT03207776/Prot_SAP_000.pdf